CLINICAL TRIAL: NCT00675870
Title: Phase II Study of NRX 195183 Therapy for Patients With Relapsed or Refractory Acute Promyelocytic Leukemia
Brief Title: Study of NRX 195183 Therapy for Patients With Relapsed or Refractory Acute Promyelocytic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NuRx Pharmaceuticals, Inc. (Industry)
Responsible Party: Roshantha A. Chandraratna, PhD, MBA, Chief Scientific Officer, NuRx Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 195183-202
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia; Cancer; Leukemia; APL; ATRA; Tretinoid; Vesanoid; Retinoic Acid Receptor Alpha; All Trans Retinoic Acid; Arsenic Trioxide; Trisenox; Retinoid; Relapsed or Refractory Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Neoplasms; Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: NRX 195183 Soft Gelatin Capsule

INTERVENTIONS:
Drug: NRX 195183 Soft Gelatin Capsule — Daily oral NRX 195183 administration for 90 days to assess CR rate. Patients with CR may continue maintenance therapy after a 2-week drug holiday. Maintenance therapy will consist of two 3-month daily oral NRX 195183 administration separated by a 2-week drug holiday.

SUMMARY:
The purpose of this study is to determine whether NRX 195183 is effective in the treatment of relapsed or refractory Acute Promyelocytic Leukemia

DETAILED DESCRIPTION:
A common current therapeutic approach to APL uses oral ATRA and chemotherapy in induction and consolidation. This approach has significantly improved survival in newly diagnosed APL patients. However, approximately 30% of patients relapse. Recently, an approach involving the combination of oral ATRA and arsenic trioxide has been tested. The prognosis for relapsed patients is very poor. This study seeks to investigate NRX 195183 monotherapy in patients who have failed or are resistant to or are intolerant of any prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of APL morphology or FAB M3 variant confirmed by RT-PCR assay or chromosome analysis/FISH showing t(15:17) translocation. Patients must also have relapse from, resistance to or intolerance of any one or more of the following therapies:

  * ATRA
  * Cytotoxic chemotherapy
  * Arsenic trioxide
* Patients must be 18 or older.
* Bilirubin equal or less than 1.5 times the upper limit of normal.
* Creatinine equal or less than 1.5 times the upper limit of normal.
* Patients entered into this study should be non-pregnant and non-nursing and should not plan on becoming pregnant while on treatment. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control. There is an extremely high risk that a severely deformed infant will result if NRX 195183 is administered during pregnancy.

Exclusion Criteria:

* Non-APL, AML patients should be excluded from the study.
* Other serious illnesses which would limit survival to 6 months.
* Psychiatric conditions which would prevent compliance with treatment or informed consent.
* Uncontrolled or severe cardiovascular disease. This would include history of a recent acute myocardial infarction, uncontrolled congestive heart failure, or active angina.
* AIDS or HIV positive patients, although HIV test is not required for accrual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Complete Remission | 90 Days

SECONDARY OUTCOMES:
Molecular Complete Remission | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States